CLINICAL TRIAL: NCT00185653
Title: Mixed Chimera Allogeneic Transplantation From Matched Unrelated Donors for the Treatment of Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Robert Lowsky, Principal Investigator, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT126; 73506; BMT126; NCT00185653
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Procedure: Autologous followed by non-myeloablative allogeneic transplantation

SUMMARY:
The purpose of the study is to determine the toxicity and feasibility of non-myeloablative allogeneic hematopoietic cell transplants for multiple myeloma from unrelated donors.

DETAILED DESCRIPTION:
The primary objective of the protocol is to evaluate the toxicity and tolerability of this mixed chimerism matched unrelated donor allogeneic transplant approach for patients with multiple myeloma. Response, toxicity, survival and graft-versus-host disease will be evaluated.

ELIGIBILITY:
Inclusion Criteria:a) Multiple myeloma which is responsive to therapy. Eligible patients may have early or relapsed disease. Patients must have Stage II-III disease or have progression after initial treatment of Stage I disease. Patients who have relapsed following autologous transplantation may be eligible for this protocol.

b) Age <= 60 years. c) No prior therapy which would preclude the use of low-dose total body irradiation.

d) Patients must have their pathology reviewed and the diagnosis confirmed at Stanford University Medical Center. Patients with smoldering multiple myeloma, monoclonal gammopathy of unknown significance, or amyloidosis will be excluded from this study.

e) Patients must have a Karnofsky performance status > 70%. f) DLCO >= 60% predicted. g) ALT and AST must be < 2X normal. Total bilirubin less than 2 mg/dl. h) Serum creatinine < 2.0 or 24-hour creatinine clearance >= 50 ml/min. i) Patients must be HIV negative. j) Pregnant or lactating women will not be eligible to participate. k) Patients must provide signed, informed consent. Exclusion Criteria:a) Severe psychological or medical illness b) Patients who have undergone prior allogeneic hematopoietic cell transplantation will not be eligible for this study.

c) Patients who have an HLA-identical sibling donor will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2000-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and laboratory-measured efficacy of mixed chimera unrelated donor allogeneic transplants.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States